CLINICAL TRIAL: NCT04013841
Title: Bowel Preparation for Left Side Colon Surgery Impact on the Intestinal Microbiome: Oral Preparation vs Enema
Brief Title: Bowel Preparation Impact on the Intestinal Microbiome: Oral Preparation vs Enema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vilnius University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Rimantas Bausys, Principle Investigator, Vilnius University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BowelPrepMicrobiome
Record Dates: First submitted 2019-07-07; First posted 2019-07-10 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Enema

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral preparation (Experimental): The bowel preparation prior to colorectal resection will be conducted using oral-agents
  Interventions: Other: Oral-agents/Enema
- Enema preparation (Experimental): The bowel preparation prior to colorectal resection will be conducted using rectal enema
  Interventions: Other: Oral-agents/Enema

INTERVENTIONS:
Other: Oral-agents/Enema — 1. Oral-agents for mechanical bowel preparation prior to left-side colorectal resection
  2. Enema for mechanical bowel preparation prior to left-side colorectal resection

SUMMARY:
Mechanical bowel preparation for left-sided colorectal surgery remains standard in most cases. However, there are some discrepancies on how to prepare the bowl, while rectal enema and oral agents are both available methods.

The knowledge of intestinal microbiome role on surgical outcomes is increasing, since few recent reports linked microbiome composition to postoperative complications, such as anastomotic insufficiency. Although, it is not clear how the bowel preparation affects the gut microbiome. Therefore, different bowel preparation techniques impact on gut microbiome will be studied.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 y.;
2. Signed informed consent;
3. Left-side colorectal resection for colorectal cancer;

Exclusion Criteria:

1. Anticipated ileostoma;
2. Allergy to oral preparation agents;
3. Multivisceral surgery;
4. Emergency surgery;
5. History of inflammatory bowel disease;
6. History of surgery disrupting gastrointestinal tract integrity;
7. Signs of tumor obturating the lumen of the bowel;
8. Pregnancy;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-08 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Intestinal microbiome composition | 6 days after surgery
  Significant differences in the beta-diversity of the intestinal microbiome between oral and enema groups

SECONDARY OUTCOMES:
Intestinal microbiome composition | 30 days after surgery
  Significant differences in the beta-diversity of the intestinal microbiome between oral and enema groups
Intestinal microbiome composition | 6 and 30 days after surgery
  Significant differences in the alpha-diversity of the intestinal microbiome between oral and enema groups

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rauduvyte K, Kazlauskaite P, Kryzauskas M, Ignatavicius P, Poskus T, Sabaliauskaite R, Mlynska A, Sestokaite A, Luksta M, Bausys R, Jakubauskas M, Bausys A. Preoperative TNF-alpha predicts uneventful postoperative outcomes in patients undergoing colorectal cancer surgery. Sci Rep. 2025 Jul 1;15(1):21878. doi: 10.1038/s41598-025-06667-6. PMID 40596170
- [Derived] Zukauskaite K, Horvath A, Gricius Z, Kvietkauskas M, Bausys B, Dulskas A, Kuliavas J, Bausys R, Letautiene SR, Vaicekauskaite I, Sabaliauskaite R, Bausys A, Stadlbauer V, Jarmalaite S. Impact of mechanical bowel preparation on the gut microbiome of patients undergoing left-sided colorectal cancer surgery: randomized clinical trial. Br J Surg. 2024 Aug 30;111(9):znae213. doi: 10.1093/bjs/znae213. PMID 39222391